CLINICAL TRIAL: NCT06245330
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Efficacy and Correlation With AKR1C3 Enzyme Expression of AST-001 in Subjects With Advanced Solid Tumors
Brief Title: A Phase I/II Study of AST-001 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascentawits Pharmaceuticals, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AT-001-001
Record Dates: First submitted 2024-01-10; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation phase (Experimental): AST-001 (5.0 mg/m^2 to 40.0 mg/m^2) will be administered by IV infusion on Days 1, 8 and 15 of each 28-day cycle to determine the MTD and RP2D with a BOIN design.
  Interventions: Drug: AST-001
- phase II pancreatic cancer (Experimental): AST-001 (RP2D) will be administered by IV infusion on Days 1, 8 and 15 of each 28-day cycle
  Interventions: Drug: AST-001

INTERVENTIONS:
Drug: AST-001 — liquid formulation for Intravenous infusion

SUMMARY:
A first-in-human open-label, Phase I/II study to evaluate the safety, tolerability, MTD/RP2D, PK, and preliminary efficacy of AST-001 administered as a single agent.

ELIGIBILITY:
* phase I: dose escalation phase

Inclusion Criteria:

1. Patient has ability to understand the risks of the study and is willing to comply with the protocol and has signed a written informed consent.
2. Aged 18-70 years (inclusive), males and females.
3. Histologically or cytologically confirmed solid malignancy that is metastatic or unresectable and for which standard curative do not exist or are no longer effective.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Expected life expectancy ≥ 12 weeks
6. Recovered from toxicities of prior therapy to Grade 0 or 1
7. An adequate renal, liver and bone marrow function.

Exclusion Criteria:

1. History of another primary malignancy within 2 years prior to Day 1, except for adequately treated basaloma, in situ cancer, or other cancers whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the current study.
2. Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1.
3. Treatment with radiation therapy, chemotherapy, biotherapy, targeted therapies or hormones within 4 weeks prior to Day 1.
4. Receiving investigational therapy within 4 weeks prior to Day 1.
5. Concomitant use of repaglinide, medium/strong CYP2C8/CYP2B6/ CYP2C9 inhibitors/inducers.
6. Pleural effusion or ascites which need to be drained every other week or more frequently.
7. HBV infection and HBV-DNA ≥ 2,000 IU/mL
8. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
9. History of human immunodeficiency virus (HIV) infection or syphilis infection.
10. History of cardiac disease fits any of the following conditions：

    1. NYHA III or IV CHF；
    2. QTcF : male > 450ms，female > 470ms；
    3. Myocardial infarction, bypass surgery, stent surgery within 6 months prior to Day 1；
    4. Other cardiac disease that the investigator judged unsuitable for inclusion.
11. Females who are pregnant or breast-feeding
12. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
13. Previously allergic to ethanol, polyoxyethylene (35) castor oil, N, N-dimethylacetamide.
14. Unwillingness or inability to comply with the study protocol for any reason

    * phase II: pancreatic cancer

Inclusion Criteria:

1. Patient has ability to understand the risks of the study and is willing to comply with the protocol and has signed a written informed consent.
2. Aged 18-70 years (inclusive), males and females.
3. Histologically or cytologically confirmed pancreatic cancer that is unresectable or cannot be controlled by local treatment and for which standard curative do not exist or are no longer effective.
4. At least one measurable lesion that meets RECIST 1.1 criteria.
5. Can provide pathological wax blocks or sections (including archived pathological wax blocks or sections) for AKR1C3 expression analysis and be confirmed that AKR1C3 expression is strongly positive.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Expected life expectancy ≥ 12 weeks
8. Recovered from toxicities of prior therapy to Grade 0 or 1
9. An adequate renal, liver and bone marrow function.

Exclusion Criteria:

1. History of another primary malignancy within 2 years prior to Day 1, except for adequately treated basaloma, in situ cancer, or other cancers whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the current study.
2. Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1.
3. Treatment with radiation therapy, chemotherapy, biotherapy, targeted therapies or hormones within 4 weeks prior to Day 1.
4. Receiving investigational therapy within 4 weeks prior to Day 1.
5. Concomitant use of repaglinide, medium/strong CYP2C8/CYP2B6/ CYP2C9 inhibitors/inducers.
6. Pleural effusion or ascites which need to be drained every other week or more frequently.
7. HBV infection and HBV-DNA ≥ 2,000 IU/mL
8. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
9. History of human immunodeficiency virus (HIV) infection or syphilis infection.
10. History of cardiac disease fits any of the following conditions：

    1. NYHA III or IV CHF；
    2. QTcF : male > 450ms，female > 470ms；
    3. Myocardial infarction, bypass surgery, stent surgery within 6 months prior to Day 1；
    4. Other cardiac disease that the investigator judged unsuitable for inclusion.
11. Females who are pregnant or breast-feeding
12. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
13. Previously allergic to ethanol, polyoxyethylene (35) castor oil, N, N-dimethylacetamide.
14. Unwillingness or inability to comply with the study protocol for any reason

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Adverse events will be noted as it occurs. Timeframe for measure begins after informed consent until 30 days after last dose of study drug.
  Adverse events will be graded according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
Assess safety changes in electrocardiogram (ECG) | Day 1 of each cycle(there are 26 cycles; 28 days for each cycle)
  Resting 12-lead ECGs will be obtained from all subjects' pre-AST-001 infusion and within 30 minutes post-AST-001 infusion in order to assess any impact AST-001 may have on the QT interval as assessed by the Fridericia's Correction Formula (QTcF).
Assess safety changes of body weight. | pre-AST-001 infusion of each cycle (there are 26 cycles; 28 days for each cycle)
  If during treatment a subject's body weight changes by >10%, the dose should be adjusted.
Number of participants with dose limiting toxicities (DLTs) | Throughout Cycle 1 (28 days for each cycle)
  A DLT is defined as the occurrence of Grade 3/4 adverse events within the first cycle (the first 28 days) of treatment that are considered by the investigator to be at least possibly related to AST-001.
Define the Recommended Phase 2 Dose (RP2D) | Days 1, 8 and 15 of each cycle (all 26 cycles and there are 28 days for each cycle)
  Determination of the MTD, based on the frequently of DLTs observed in Cycle 1 in subjects recruited to the Dose Escalation Phase.
Pharmacokinetics (PK) - Time to maximum concentration (Tmax) | Days 1 and 15 of Cycle 1 (first cycle of 26 cycles and there are 28 days for each cycle)
  Tmax of AST-001 and AST-2660 will be computed for each subject where possible
PK - Maximum peak plasma concentration (Cmax) | Days 1 and 15 of Cycle 1 (first cycle of 26 cycles and there are 28 days for each cycle)
  Cmax of AST-001 and AST-2660 will be computed for each subject where possible.
PK - Area under the concentration-time curve (AUClast) PK - Area under the concentration-time curve (AUClast) | Days 1 and 15 of Cycle 1 (first cycle of 26 cycles and there are 28 days for each cycle)
  AUClast from Hour 0 through the last quantifiable concentration time (LQCT), where LQCT is the time at which the last sample with a quantifiable concentration was drawn
PK - Half-life (T1/2) | Days 1 and 15 of Cycle 1 (first cycle of 26 cycles and there are 28 days for each cycle)
  T1/2 computed as ln (2)/Kel of AST-001 and AST-2660 will be computed for each subject where possible.
Efficacy: Objective response rate(ORR) | up to 26 cycles (there are 28 days for each cycle)
  ORR will be assessed as a primary outcome in phase II.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, Principal Investigator — Study Principal Investigator
Locations (1):
- Jinlin Cancer Hospital, Changchun, Jinlin, China